CLINICAL TRIAL: NCT00407927
Title: A Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Safety, Efficacy, and Tolerability Study of Two Doses of Epinastine Nasal Spray (0.05% and 0.1%) vs. Placebo in Subjects With Seasonal Allergic Rhinitis
Brief Title: A Study of Epinastine Nasal Spray in Subjects With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 033-101
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

INTERVENTIONS:
Drug: Epinastine Nasal Spray

SUMMARY:
The purpose of this trial is to determine the safety, efficacy and tolerability of two doses of the study drug compared to placebo for the treatment of subjects with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* A documented history of seasonal allergic rhinitis to mountain cedar pollen

Exclusion Criteria:

* Significant medical condition
* Cardiovascular abnormality
* Have a significant physical obstruction in the nose
* Started or had a change in immunotherapy within the 30 days prior to

screening

* Have nasal ulceration(s) or any active nasal bleeding
* Require use of allergy medications during the study
* Require use of asthma medications other than as needed albuterol

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in nasal symptom scores

SECONDARY OUTCOMES:
Change in non-nasal symptom scores and quality of life scores
Standard safety assessments

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Allergy & Asthma Associates, Austin, Texas
  - Lovelace Scientific Resources, Inc., Austin, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas